CLINICAL TRIAL: NCT00105729
Title: Substance Abuse Self-Help Group Referral: Outcome and Services Use
Brief Title: Substance Abuse Self-Help Group Referral: Outcomes and Services Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIR 20-067
Record Dates: First submitted 2005-03-16; First posted 2005-03-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2006-09

CONDITIONS: Substance Use Disorders
Keywords: Self-help groups; Referral and consultation
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Intensive referral to 12-step self-help groups

INTERVENTIONS:
Behavioral: Intensive referral to 12-step self-help groups

SUMMARY:
Self-help groups (SHGs) have become an important component of the system of care for patients with substance use disorders (SUDs). SUD patients' participation in SHGs has been linked to lower relapse rates and less use of additional treatment services.

DETAILED DESCRIPTION:
Background:

Self-help groups (SHGs) have become an important component of the system of care for patients with substance use disorders (SUDs). SUD patients' participation in SHGs has been linked to lower relapse rates and less use of additional treatment services.

Objectives:

The first objective was to implement and validate procedures to help counselors make effective referrals to SHGs for SUD patients. This project randomly assigned SUD outpatients to a standard referral or an intensive referral condition. We are determining the extent to which intensive referral increased patients' SHG attendance and involvement in comparison to standard referral. The second objective is to determine whether patients who received intensive referral to SHGs have better substance use and functioning outcomes over the 1-year follow-up period, and less use of formal treatment services, thereby reducing costs for VA, than those who received standard referral. The long-term goal is to develop and implement guidelines to facilitate SUD patients' participation in SHGs and thereby improve their quality of life and decrease their use of VA's specialized SUD treatment services.

Methods:

This project used a randomized design in which 345 patients entering VA outpatient SUD treatment were randomly assigned to either standard or intensive referral to SHGs. Standard referral consisted of the counselor recommending SHG participation. The keys to intensive referral included the counselor facilitating direct contact between the patient and a member of the SHG, and counselor follow-up on the recommendation for self-help. Patients were followed at 6 months and 1 year to determine whether intensive referral resulted in more self-help attendance and involvement; in better substance use and functioning outcomes (using the Addiction Severity Index); and in less use of VA services and lower treatment costs (using methods of the VA Health Economics Resource Center). To make these determinations, we are conducting analyses at each follow-up, and then will use hierarchical linear modeling to examine the benefits of intensive referral over time.

Status:

Project work is ongoing.

ELIGIBILITY:
Inclusion Criteria:

Consecutive substance use disorder outpatients at VA PA HCS and is not cognitively impaired.

Exclusion Criteria:

Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Estimated)
Dates: Start 2003-01; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
DRUG USE AND ALCOHOL USE AT 6 MONTHS AND 1 YEAR

SECONDARY OUTCOMES:
SUBSTANCE ABUSE AND PSYCHIATRIC SERVICES USE AT 6 MONTHS AND 1 YEAR

CONTACTS AND LOCATIONS:
Overall Officials: Christine Timko, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

REFERENCES:
- [Result] Timko C, Billow R, DeBenedetti A. Determinants of 12-step group affiliation and moderators of the affiliation-abstinence relationship. Drug Alcohol Depend. 2006 Jun 28;83(2):111-21. doi: 10.1016/j.drugalcdep.2005.11.005. Epub 2005 Dec 9. PMID 16338102
- [Result] Timko C, DeBenedetti A. A randomized controlled trial of intensive referral to 12-step self-help groups: one-year outcomes. Drug Alcohol Depend. 2007 Oct 8;90(2-3):270-9. doi: 10.1016/j.drugalcdep.2007.04.007. Epub 2007 May 24. PMID 17524574